CLINICAL TRIAL: NCT02407457
Title: Multicenter, Post-Market Study to Assess Outcomes of Patients Treated With the AFX System Compared to Other EVAR Devices for Endovascular Abdominal Aortic Aneurysm Repair: LEOPARD
Brief Title: Post-Market Study to Assess Outcomes of Patients Treated With AFX System Compared to Other EVAR Devices
Acronym: LEOPARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-0011
Record Dates: First submitted 2015-03-06; First posted 2015-04-03 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AFX EVAR AAA Graft System (Active Comparator): Subjects randomized to receive the Endologix AFX Endovascular Graft System for implantation to repair Abdominal Aortic Aneurysm via femoral access.
  Interventions: Device: AFX EVAR AAA Graft System
- FDA Approved EVAR AAA Graft Systems (Active Comparator): Subjects randomized to receive the comparator AAA Endovascular Graft System for implantation to repair Abdominal Aortic Aneurysm via femoral access.
  Interventions: Device: FDA Approved EVAR AAA Graft Systems

INTERVENTIONS:
Device: AFX EVAR AAA Graft System — Endvovascular Abdominal Aneurysm Repair (EVAR) using commerically available, FDA approved endovascular graft systems implanted via femoral access.
  Arms: AFX EVAR AAA Graft System
Device: FDA Approved EVAR AAA Graft Systems
  Arms: FDA Approved EVAR AAA Graft Systems

SUMMARY:
The objective of this post-market trial is to evaluate Endologix AFX endovascular AAA system with anatomical fixation against other approved Endovascular systems with proximal fixation. Multiple U.S clinical centers will be involved in the trial to include a broad range of experience. Imaging data will be evaluated by an independent core lab.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, multi-center trial, intended to evaluate the outcomes of contemporary EVAR (Endovascular Aneurysm Repair) in a real world population. The trial is designed to compare the anatomically stabilized AFX Endograft System to a reference group of proximally fixated EVAR devices. Patients will be randomized between the two groups.

Randomization will be 1:1. Each investigator will select one comparator device of their choice before enrolling the first patient. The study will sequentially evaluate non-inferiority and superiority hypotheses.

Up to 80 sites with experience in EVAR and up to 800 subjects will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old
2. Subjects with minimum of 2 year life expectancy
3. Subjects have signed the informed consent document for data release
4. Subjects with infrarenal AAA who are assessed by the Investigator to be eligible for endovascular Abdominal Aortic Aneurysm Repair with the trial devices.

Exclusion Criteria:

1. Currently participating in another study where primary endpoint has not been reached yet
2. Known allergy to any of the device components
3. Pregnant (females of childbearing potential only)
4. Subjects with pre-existing EVAR, e.e. in need of repair/intervention of a previously failed EVAR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kwolek, MD, Principal Investigator — Endologix
Locations (56):
- United States (56):
  - Eliza Coffee Medical Center, Florence, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Carondelet Heart and Vascular Institute, Tucson, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Long Beach VA Hospital, Long Beach, California
  - Sacramento Vascular Sugeons, Sacramento, California
  - Kaiser - Santa Clara, Santa Clara, California
  - Penrose St. Francis Health, Colorado Springs, Colorado
  - Hartford Hospital, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Mayo Jacksonville, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Vascular Institute of Central Florida, Orlando, Florida
  - Sarasota Vascular Specialists, Sarasota, Florida
  - USF/Tampa VA, Tampa, Florida
  - Emory/Grady, Atlanta, Georgia
  - Navicent Health Medical Center, Macon, Georgia
  - Peachtree Vascular Specialists, Stockbridge, Georgia
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Cadence Physician Group, Winfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Franciscan - St. Francis Hospital, Indianapolis, Indiana
  - University of Iowa Healthcare, Iowa City, Iowa
  - The Iowa Clinic Cardiovascular Services, West Des Moines, Iowa
  - Surgical Care Associates, Louisville, Kentucky
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Baton Rouge Vascular Specialty Center, Baton Rouge, Louisiana
  - VA Maryland Health Care System, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - North MS Medical Center, Tupelo, Mississippi
  - University of Missouri, Columbia, Missouri
  - Kansas City Vascular, North Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - The Vascular Group, Albany, New York
  - VA Western New York Healthcare System, Buffalo, New York
  - Wake Forest, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Innovation Center, Kettering Health Network, Kettering, Ohio
  - Neo Vascular (Lake West), Willoughby, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - North Central Heart, Sioux Falls, South Dakota
  - Cardiothoracic & Vascular Surgeons, Austin, Texas
  - University of Texas Health, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Peacehealth Southwest Medical Center, Vancouver, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Prinssen M, Verhoeven EL, Buth J, Cuypers PW, van Sambeek MR, Balm R, Buskens E, Grobbee DE, Blankensteijn JD; Dutch Randomized Endovascular Aneurysm Management (DREAM)Trial Group. A randomized trial comparing conventional and endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2004 Oct 14;351(16):1607-18. doi: 10.1056/NEJMoa042002. PMID 15483279
- [Background] Volodos' NL, Karpovich IP, Shekhanin VE, Troian VI, Iakovenko LF. [A case of distant transfemoral endoprosthesis of the thoracic artery using a self-fixing synthetic prosthesis in traumatic aneurysm]. Grudn Khir. 1988 Nov-Dec;(6):84-6. No abstract available. Russian. PMID 3220297
- [Background] Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG; EVAR trial participants. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet. 2004 Sep 4-10;364(9437):843-8. doi: 10.1016/S0140-6736(04)16979-1. PMID 15351191
- [Background] Brown LC, Greenhalgh RM, Thompson SG, Powell JT; EVAR Trial Participants. Does EVAR alter the rate of cardiovascular events in patients with abdominal aortic aneurysm considered unfit for open repair? Results from the randomised EVAR trial 2. Eur J Vasc Endovasc Surg. 2010 Apr;39(4):396-402. doi: 10.1016/j.ejvs.2010.01.002. Epub 2010 Jan 21. PMID 20096611
- [Background] Stroupe KT, Lederle FA, Matsumura JS, Kyriakides TC, Jonk YC, Ge L, Freischlag JA; Open Versus Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Cost-effectiveness of open versus endovascular repair of abdominal aortic aneurysm in the OVER trial. J Vasc Surg. 2012 Oct;56(4):901-9.e2. doi: 10.1016/j.jvs.2012.01.086. Epub 2012 May 27. PMID 22640466
- [Background] De Bruin JL, Baas AF, Buth J, Prinssen M, Verhoeven EL, Cuypers PW, van Sambeek MR, Balm R, Grobbee DE, Blankensteijn JD; DREAM Study Group. Long-term outcome of open or endovascular repair of abdominal aortic aneurysm. N Engl J Med. 2010 May 20;362(20):1881-9. doi: 10.1056/NEJMoa0909499. PMID 20484396
- [Derived] Kwolek CJ, Ouriel K, Stucky FS, Rao VK, Pons PJ, Wilson SE, Kujath SW. Five-year results of the LEOPARD trial of commercially available endografts. J Vasc Surg. 2023 Aug;78(2):324-332.e2. doi: 10.1016/j.jvs.2023.04.011. Epub 2023 Apr 15. PMID 37068528

RESULTS

PARTICIPANT FLOW:
Groups:
- FDA Approved EVAR AAA Graft Systems: Subjects randomized to receive the comparator AAA Endovascular Graft System for implantation to repair Abdominal Aortic Aneurysm via femoral access.
  FDA Approved EVAR AAA Graft Systems
Period: Baseline
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 235 | 220
Completed | 235 | 220
Not Completed | 0 | 0
Period: 1 Month
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 235 | 220
Completed | 229 | 214
Not Completed | 6 | 6
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — missed visit | 2 | 5
Period: 6-Month
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 231 | 219
Completed | 211 | 194
Not Completed | 20 | 25
Not completed — Death | 2 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — missed visit | 16 | 14
Not completed — Open Repair | 0 | 1
Period: 1 Year
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 227 | 208
Completed | 194 | 180
Not Completed | 33 | 28
Not completed — Death | 6 | 11
Not completed — Lost to Follow-up | 3 | 2
Not completed — Missed Visit | 24 | 14
Not completed — Open Repair | 0 | 1
Period: 2-year
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 218 | 194
Completed | 184 | 159
Not Completed | 34 | 35
Not completed — Death | 14 | 8
Not completed — Lost to Follow-up | 7 | 10
Not completed — Missed Visit | 13 | 15
Not completed — Open Repair | 0 | 2
Period: 3-year
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 197 | 174
Completed | 158 | 138
Not Completed | 39 | 36
Not completed — Death | 11 | 10
Not completed — Lost to Follow-up | 9 | 10
Not completed — Missed Visit | 19 | 16
Period: 4-year
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 177 | 133
Completed | 131 | 95
Not Completed | 46 | 38
Not completed — Death | 18 | 10
Not completed — Lost to Follow-up | 10 | 12
Not completed — Missed Visit | 18 | 16
Period: 5-year
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Started | 148 | 131
Completed | 107 (Due to the time frame of the study - subjects have not passed 5-year.) | 114
Not Completed | 41 | 17
Not completed — Death | 10 | 3
Not completed — Lost to Follow-up | 22 | 13
Not completed — Missed Visit | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems | Total
Number analyzed (Participants) | 235 | 220 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8) | 72 (8) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 212 | 192 | 404
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 225 | 199 | 424
  Non-caucasian | 10 | 21 | 31
ASA Classification [Count of Participants; unit: Participants] — The first row (ASA Class 1 / 2) reflects patients with fewer health concerns and the second row (Class 3/4/5), reflects patients with more severe medical co-morbidities. **Note, this data reflects counts of participants, not frequency.
  Participants
    ASA Class 1/2 | 71 | 62 | 133
    ASA Class 3/4/5 | 164 | 158 | 322

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Absence of Aneurysm Related Complications (ARC)
Description: ARC is a composite of the most relevant EVAR outcomes and includes:
  * Peri-Operative Death (< 30 days)
  * Rupture
  * Conversion to OSR
  * Endoleaks; post-operative
  * Migration (≥ 10mm)
  * Aneurysm Enlargement (≥ 5mm)
  * Endograft Limb Occlusions
  * Reinterventions for device- or aneurysm-related complications
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants | 195 | 175

2. Secondary Outcome: The Number of MAEs
Description: Major Adverse Events
Time Frame: At 30 days, 12 months, and annually up to five years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  Bleeding : 30 days | 3 | 4
  Bleeding : 12 Months | 3 | 4
  Bleeding : 24 Months | 0 | 0
  Bleeding : 36 Months | 0 | 0
  Bleeding : 48 Months | 1 | 1
  Bleeding : 60 Months | 0 | 0
  Cardiac : 30 days | 4 | 1
  Cardiac : 12 Months | 5 | 12
  Cardiac : 24 Months | 2 | 2
  Cardiac : 36 Months | 6 | 4
  Cardiac : 48 Months | 9 | 0
  Cardiac : 60 Months | 4 | 2
  GI : 30 days | 1 | 0
  GI : 12 Months | 1 | 0
  GI : 24 Months | 0 | 0
  GI : 36 Months | 0 | 0
  GI : 48 Months | 0 | 0
  GI : 60 Months | 0 | 0
  Malignancies : 30 days | 1 | 0
  Malignancies : 12 Months | 4 | 5
  Malignancies : 24 Months | 5 | 3
  Malignancies : 36 Months | 1 | 1
  Malignancies : 48 Months | 2 | 0
  Malignancies : 60 Months | 2 | 1
  Miscellaneous : 30 days | 2 | 0
  Miscellaneous : 12 Months | 5 | 2
  Miscellaneous : 24 Months | 1 | 0
  Miscellaneous : 36 Months | 3 | 6
  Miscellaneous : 48 Months | 0 | 5
  Miscellaneous : 60 Months | 3 | 1
  Neurological : 30 days | 1 | 0
  Neurological : 12 Months | 2 | 4
  Neurological : 24 Months | 6 | 3
  Neurological : 36 Months | 5 | 2
  Neurological : 48 Months | 2 | 1
  Neurological : 60 Months | 1 | 2
  Pulmonary : 30 days | 1 | 0
  Pulmonary : 12 Months | 2 | 3
  Pulmonary : 24 Months | 5 | 2
  Pulmonary : 36 Months | 0 | 2
  Pulmonary : 48 Months | 2 | 3
  Pulmonary : 60 Months | 3 | 1
  Renal : 30 days | 0 | 0
  Renal : 12 Months | 1 | 4
  Renal : 24 Months | 0 | 0
  Renal : 36 Months | 0 | 0
  Renal : 48 Months | 0 | 0
  Renal : 60 Months | 0 | 0
  Wound : 30 days | 0 | 0
  Wound : 12 Months | 0 | 1
  Wound : 24 Months | 0 | 0
  Wound : 36 Months | 0 | 0
  Wound : 48 Months | 0 | 0
  Wound : 60 Months | 0 | 0
  Vascular : 30 days | 0 | 0
  Vascular : 12 Months | 0 | 0
  Vascular : 24 Months | 0 | 0
  Vascular : 36 Months | 1 | 0
  Vascular : 48 Months | 2 | 0
  Vascular : 60 Months | 0 | 0

3. Secondary Outcome: The Number of Participants With Aneurysm Related Complications (ARC)
Description: ARC is a composite outcome
Time Frame: Post 12 Months up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 52 | 64
  24 Months | 23 | 29
  36 Months | 22 | 22
  48 Months | 23 | 16
  60 Months | 19 | 16

4. Secondary Outcome: The Number of Participants With Aneurysm Related Mortality
Description: Death related to the aneurysm
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  1 Year | 3 | 1
  2 Years | 0 | 1
  3 Years | 1 | 1
  4 Years | 2 | 1
  5 Years | 0 | 0

5. Secondary Outcome: Number of Type Ia Endoleaks
Description: Number of participants with Type Ia endoleaks at 12 months, 24 months, 36 months, 48 months and 60 months. Type Ia endoleak defined as persistent leak around the top of the stent graft identified during imaging surveillance at the different timepoints.
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 2 | 0
  24 Months | 0 | 0
  36 Months | 0 | 1
  48 Months | 3 | 1
  60 Months | 0 | 1

6. Secondary Outcome: Number of Type Ib Endoleaks
Description: Number of participants with Type Ib endoleaks at 12 months, 24 months, 36 months, 48 months and 60 months. Type Ib endoleak defined as persistent leak around the bottom of the stent graft identified during imaging surveillance at the different timepoints.
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 4 | 3
  24 Months | 0 | 0
  36 Months | 0 | 0
  48 Months | 0 | 0
  60 Months | 1 | 1

7. Secondary Outcome: Number Endoleaks Type II
Description: Number of participants with Type II endoleaks at 12 months, 24 months, 36 months, 48 months and 60 months. Type II endoleak defined as persistent blood flow into the aneurysm sac from branches of the aorta identified during imaging surveillance at the different timepoints.
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 36 | 48
  24 Months | 5 | 3
  36 Months | 2 | 4
  48 Months | 1 | 0
  60 Months | 0 | 3

8. Secondary Outcome: Number of Endoleaks Type IIIa
Description: Number of participants with Type IIIa endoleaks at 12 months, 24 months, 36 months, 48 months and 60 months. Type IIIa endoleak defined as persistent leak from the overlapping parts of the stent graft identified during imaging surveillance at the different timepoints.
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 0 | 0
  24 Months | 0 | 0
  36 Months | 0 | 0
  48 Months | 0 | 0
  60 Months | 1 | 0

9. Secondary Outcome: Number of Endoleaks Type IIIb
Description: Number of participants with Type IIIb endoleaks at 12 months, 24 months, 36 months, 48 months and 60 months. Type IIIb endoleak defined as persistent leak as a consequence of graft rupture, identified during imaging surveillance at the different timepoints.
Time Frame: Up to Five Years
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 0 | 0
  24 Months | 0 | 0
  36 Months | 1 | 0
  48 Months | 0 | 0
  60 Months | 0 | 0

10. Secondary Outcome: Number of Participants With Aneurysm Rupture
Description: Number of Participants with Aneurysm Rupture at 12 Months, 24 Months, 36 Months, 48 Months and 60 Months
Time Frame: 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 0 | 0
  24 Months | 0 | 0
  36 Months | 1 | 0
  48 Months | 1 | 1
  60 Months | 0 | 0

11. Secondary Outcome: Number of Participants With Open Conversion
Description: Number of Participants that underwent an Open Conversions at 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Time Frame: 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 0 | 3
  24 Months | 0 | 1
  36 Months | 0 | 0
  48 Months | 0 | 0
  60 Months | 0 | 0

12. Secondary Outcome: Number of Participants With Aneurysm Expansion
Description: Number of Participants with Aneurysm Expansion at 12 Months, 24 Months, 36 Months, 48 months, 60 Months
Time Frame: 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 2 | 4
  24 Months | 4 | 1
  36 Months | 2 | 3
  48 Months | 9 | 4
  60 Months | 7 | 5

13. Secondary Outcome: Number of Patients With Endograft Occlusion
Description: Number of Patients with Endograft Occlusion at 12 Months, 24 Months, 36 Months, 48 Months and 60 Months
Time Frame: 12 Months, 24 Months, 36 Months, 48 Months and 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  12 Months | 3 | 8
  24 Months | 0 | 1
  36 Months | 0 | 1
  48 Months | 1 | 1
  60 Months | 1 | 0

14. Secondary Outcome: Number of Participants With Device-Related Secondary Interventions
Description: Number of Participants with Device-Related Secondary Interventions at 30 days, 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Time Frame: 30 days, 12 Months, 24 Months, 36 Months, 48 Months, 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants
  30 Days | 5 | 2
  12 Months | 11 | 12
  24 Months | 3 | 3
  36 Months | 7 | 4
  48 Months | 5 | 6
  60 Months | 5 | 5

15. Secondary Outcome: Number of Patients With Adjunctive Procedures
Description: Number of patients with adjunctive procedure during the implant
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
Number analyzed (Participants) | 235 | 220
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: AEs are collected through 5 year follow-up visit.
Arm/Group | AFX EVAR AAA Graft System | FDA Approved EVAR AAA Graft Systems
All-Cause Mortality (participants affected / at risk) | 64/235 | 50/220
Serious Adverse Events (participants affected / at risk) | 150/376 | 136/358
Other Adverse Events (participants affected / at risk) | 167/235 | 162/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFX EVAR AAA Graft System (N=376) | FDA Approved EVAR AAA Graft Systems (N=358)
Aneurysm Rupture (Vascular disorders) | 0 (0) | 0 (0)
cardiac (Cardiac disorders) | 52 (68) | 38 (62)
Bleeding (Blood and lymphatic system disorders) | 15 (17) | 18 (21)
Device (Vascular disorders) | 28 (34) | 22 (28)
GI (Gastrointestinal disorders) | 14 (15) | 14 (17)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 (33) | 20 (21)
neurological (Nervous system disorders) | 20 (29) | 21 (21)
pulmonary (Respiratory, thoracic and mediastinal disorders) | 37 (53) | 28 (46)
Renal (Renal and urinary disorders) | 13 (13) | 19 (20)
Vascular (Vascular disorders) | 26 (35) | 32 (40)
Wound (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (8)
Miscellaneous (General disorders) | 44 (61) | 54 (66)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFX EVAR AAA Graft System (N=235) | FDA Approved EVAR AAA Graft Systems (N=220)
Bleeding (Blood and lymphatic system disorders) | 21 (23) | 19 (22)
Cardiac (Cardiac disorders) | 52 (68) | 38 (62)
Device (Vascular disorders) | 61 (67) | 63 (72)
GI (Gastrointestinal disorders) | 14 (15) | 14 (17)
miscellaneous (General disorders) | 46 (63) | 56 (68)
Neurological (Nervous system disorders) | 22 (32) | 22 (22)
Renal (Renal and urinary disorders) | 16 (18) | 22 (23)
vascular (Vascular disorders) | 39 (51) | 44 (58)
wound (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (9)
Urogenital (Renal and urinary disorders) | 12 (14) | 9 (9)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 37 (53) | 28 (46)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 (33) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall be free to publish Institution's data/results from the Clinical Study at time of multicenter results published, notification that publication is not planned, or 18 months after the study conclusion at all centers, whichever occurs first.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT02407457/Prot_SAP_002.pdf